CLINICAL TRIAL: NCT07070154
Title: Evaluating the Efficacy of a Text Messaging-based Shisha Smoking Cessation Intervention for Young Adults in Hong Kong: A Randomised Controlled Pilot Trial
Brief Title: Evaluating the Efficacy of a Text Messaging-based Shisha Smoking Cessation Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Johnson Kai Chun LAW, Mr, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SSCI-E
Record Dates: First submitted 2025-06-18; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Intervention; Control
Keywords: shisha smoking; text-messaging based; cessation intervention; mHealth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive smartphone text messaging-based intervention and support that contained personalised messages with both text and visual elements over 6 weeks under a manualised programme. The contents of the messages within the intervention is developed based on the results of a Delphi study that identified 32 behaviour change techniques by 46 tobacco/ substance use control policy experts and mental health professionals in Hong Kong.
  Interventions: Behavioral: text-messaging based intervention
- Control (No Intervention): Participants in the control group will only receive a leaflet about the health risks of shisha smoking in either Chinese or English. The information of the leaflet will be with the exact identical contents on the leaflet received by the participants in the intervention group at Session 2.

INTERVENTIONS:
Behavioral: text-messaging based intervention — The 6-week, culture specific, text-messaging based cessation intervention for young adults in Hong Kong consists of 6 sessions: 1) Programme overview, 2) Psychoeducation on the health risks, 3) Social support, 4) Stress management, 5) Craving and withdrawal symptoms management, and 6) Summary and relapse prevention.
  Arms: Intervention

SUMMARY:
The goal of this study is to evaluate the efficacy of a culture specific text-messaging based shisha smoking cessation intervention for young adults in Hong Kong. Participants in the intervention group will receive smartphone text messaging-based intervention and support that contained personalised messages with both text and visual elements over 6 weeks under a manualised programme. Participants in the control group will only receive a leaflet about the health risks of shisha smoking (the exact identical contents received by the participants in the intervention group at a session).

All participants will complete a self-administered questionnaire at baseline, 6th- and 12th-week on their self-reported shisha abstinences, knowledge on risk, readiness to quit and attitudes on shisha smoking

DETAILED DESCRIPTION:
Shisha smoking becomes the most prevalent form of tobacco use among university students in Hong Kong. The World Health Organisation (WHO) has urged healthcare professionals, policy makers and researchers to establish cultural-specific preventing and controlling strategies for shisha smoking to address this uprising public health threat. To date, only limited researches have been conducted focusing on reducing shisha use. Medications, like varenicline and bupropion, do not outweigh behavioural intervention alone for shisha smoking cessation. Early interventions adopting from traditional tobacco smoking cessation interventions were unsuccessful in lowering the smoking rates since these interventions were unable to cover the unique features of shisha smoking, such as the social dimension, the intermittent smoking patterns and the positive attitudes towards shisha. Though a Cochrane review and meta- analysis conducted in 2022 supported the use of behavioural intervention to promote shisha abstinence (risk ratio = 3.19, 95% CI: 2.17-4.69), the level of evidence remained unsatisfactory as there were only 9 interventional studies included. The authors further suggested that more interventional studies with the use of e-health behavioural interventions for shisha smoking cessation might enhance the robustness on its efficacies.

There are strong cultural differences for the practice of shisha smoking. For example, shisha smoking is a religiously acceptable culture that deeply ingrained in Middle Eastern countries whereas it is more of a social activity in Hong Kong. In fact, culture-based shisha cessation strategies showed preliminary promising results in reducing shisha smoking. For instance, an Iranian study which recruited 212 shisha-exclusive women to evaluate the effectiveness of a 4-month in-person educational program revealed that the programme had significantly increased shisha abstinence rates, health knowledge, self-efficacy, and intention to quit when compared to the control group. A recent randomised controlled trial adopting a 6-week smoker-tailored mobile messaging intervention among 319 young adults in the US demonstrated promising results in shisha abstinence and reduced the frequency of use last up to 6 months. Up-to-date, there is no Chinese- or Hong Kong-culture based shisha smoking intervention programme available. Thus, the development of a culture specific shisha cessation interventional program for shisha smokers in Hong Kong is deemed necessary.

In short, shisha smoking is common in Hong Kong especially among youth and young adults despite its hazardous effects being similar to cigarette smoking. A growing amount of evidence has supported the use of shisha-specific behavioural interventions to address this public health threat. With the recommendation from WHO on the culture specific interventions for shisha smoking cessation but a lack of such cessation intervention in the East Asian region, there is an utmost urgent need to develop and research on a shisha smoking cessation intervention for young adults in Hong Kong.

In light of such contexts, we developed a culture specific smartphone text messaging-based shisha smoking cessation intervention for young adults in Hong Kong using the well-structured intervention mapping method. Intervention mapping is an iterative process that is commonly used to develop, implement and evaluate theory-based health or behavioural interventions. It has been widely adopted to design and implement behavioural interventions in shisha smoking and cigarette smoking cessation studies. Based on the shisha smoker's individual characteristics, the developed text messaging-based intervention contains personalised messages with both text and visual elements emphasising the negative impacts of shisha smoking. Supported by previous overseas and local studies using mHealth intervention, together with the high penetration rates of smartphone use in Hong Kong and the openness to mobile health interventions, smartphone instant messaging applications, such as WhatsApp, Telegram and Signal, will be the powerful and effective delivery modes for this text messaging-based shisha smoking cessation intervention among Hong Kong young adults.

The current randomised controlled pilot trial aims to evaluate the efficacy of the culture specific text-messaging based shisha smoking cessation intervention for young adults in Hong Kong. It is hypothesised that participants randomly allocated to the intervention can achieve higher shisha abstinence, which maintain through the three months follow-up study period than the participants in the control group. For secondary outcomes, it is hypothesised that participants in the intervention group will have lowered level of dependency, increased knowledge on risk, improved readiness to quit, and more negative attitudes on shisha smoking during the study period.

Methods Design This study will be a 3-month, prospective, 2-arm, randomised controlled pilot trial. Participants will be assessed in three timepoints: baseline, 6th-, and 12th- week. The proposed study duration will be 2 years starting from 1st December, 2024 to 30th November, 2026. The trial will be conducted in accordance with the Good Clinical Practice and the CONSORT eHealth checklist.

The newly systematically developed smartphone text-messaging based shisha smoking cessation intervention targeted for young adults in Hong Kong has never been tested. The uncertainties such as shisha smokers' acceptability and usability, or the feasibility of the intervention should be examine using a smaller sample size before scaling up to a full trial. Therefore, the current study aimed to evaluate the intervention as a pilot study.

Randomisation and blinding Consented participants will be randomised into either the intervention or the control group on a 1:1 ratio, according to the sequences from the computer-generated random number by a researcher who is independent from the recruitment and the delivery of the intervention. Allocation concealment will be performed using sealed opaque envelopes with a card inside outlining the group allocation. As shisha smoking is often a social activity, if a group of shisha smokers are recruited at the same time, the whole group will be allocated to the same treatment group to minimise the spill-over effect between the two treatment arms.

Single-blind design will be adopted for this study. To achieve effective blinding, only the outcome assessors will be blinded to the treatment arms. Blinding will not be applied to the researcher who is responsible to delivers the interventions for the two treatment arms. Though consented participants will be strongly advised not to discuss their interventions allocated between themselves, full blinding will not be employed to the participants in this study. This is because shisha is often a social activity, hence participants might still have a chance to communicate with each other, leading to the potential observational bias on the study results.

Participants A convenience sample of 100 young adult shisha smokers in Hong Kong will be recruited through local universities' email invitations, snowballing from the recruited participants and outreaching to high prevalent areas that young people smoke shisha. With references to a similar 3-month pilot randomised controlled trial in the UK that had 67 young adult shisha smokers completed the study, and assuming 30% drop-out rate, 100 young adult shisha smokers shall be appropriate to evaluate the efficacy of this novel smartphone text-messaging based intervention in this pilot study.

Procedures After eligible participants completing the informed consents and baseline assessments, they will be randomly allocated into either the intervention or the control group. For the intervention group, except for the first face-to-face encountering with the participants for informed consents and baseline assessments. The researcher will follow the intervention manual and deliver the relevant customised information and personalised messages (in Chinese or English) to the participants via their preferred smartphone text- messaging applications, such as WhatsApp, WeChat, Signal, etc. commencing on every preceding Thursday (2 days before weekend). All intervention sessions will be delivered by a researcher who will be provided with a 1-day training workshop and will be assessed by the research team before implementing the intervention. Weekly meeting will be held with the research team to monitor the progress to ensure treatment integrity and to ensure the single-blinding nature of this study. For the control group, except for the first face-to-face encountering with the participants for informed consents and baseline assessments, the researcher will only provide a leaflet about the health risks of shisha smoking in either Chinese or English to them.

Both groups will be followed-up for 3 months. Outcome assessments and data will be collected from all participants at baseline, 6th-, and 12th-week follow-up via telephone call or face-to-face interview in a research room at the University of Hong Kong. The assessments will include a self-administered (or self- reported) questionnaire booklet, and the structured interview using the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, fifth version (SCID-5). Each assessment takes around 30 minutes.

Statistical Analyses Data entry and analyses will be performed using IBM Statistical Package for the Social Sciences (SPSS), with a significance of p = 0.05. Intention to treat analysis will be adopted in this trial, missing data will be handled by the last observation carried forward approach from the 6th week follow-up onwards.

Baseline demographic characteristics, treatment adherence rate, shisha smoking, and other tobacco product smoking behaviours will be summarised with descriptive statistics in overall and by treatment condition. Between group differences will be compared by nonparametric tests, such as Pearson's chi-squared and likelihood ratio tests at baseline.

Generalised linear mixed models will be performed to explore the comparisons within and between treatment conditions for all outcome measures, including the percentage of participants who achieves shisha abstinence, the average days and smoking session (1-hour per session), frequency and duration of shisha smoking, and the mean scores and standard deviations from risk knowledges, attitudes towards shisha smoking, CL and SCID-5. Cox regression model will be conducted to determine the between group abstinence duration by hazard ratio.

ELIGIBILITY:
Inclusion Criteria:

* young adults aged 18 to 35 years who are interested in quitting shisha
* smoked shisha within the 30 days at the time of enrolment (current smoker)
* smoked for more than twelve times in 12 months (i.e., on a monthly basis)22
* able to read and communicate in Chinese or English
* agree to utilise his/her own personal mobile or smartphone to send and receive messages

Exclusion Criteria:

* scored 10 (''have already quitted'') on Contemplation Ladder assessment at baseline
* unable to provide consent
* unable to read and communicate in Chinese or English

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
shisha abstinences | From enrollment, 6-week (after treatment) and 12-week follow-up
  To compare the self-reported shisha abstinences between intervention and control group to evaluate the efficacy of the culture specific text-messaging based shisha smoking cessation intervention. Shisha abstinence is determined by self-reported last use 1) in the past 7 days using the Timeline Followback Method for active use, 2) in the past 30 days to determine current use, and 3) in the past 90 days to determine early remission in accordance with the criteria from the Diagnostic and Statistical Manual for Mental Disorders, 5th Edition.

SECONDARY OUTCOMES:
Level of dependency | From enrolment, 6-week (after treatment) and 12-week follow-up
  To compare the level of dependency between participants in intervention and control group during the study by using the diagnostic criteria from the Diagnostic and Statistical Manual of Mental Disorders, fifth version on Other Substance Use Disorder under Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, fifth version. Participants will be classified as having no (0-1), mild (2-3), moderate (4-5), or severe (6-11) substance (shisha) use disorder. The minimum score ranged from 0 to 11.
Knowledge on risk | From enrolment, 6-week (after treatment) and 12-week follow-up
  To compare the knowledge on risk between participants in intervention and control group during the study period by using a self-designed 10-item multiple choice questions (True/ False/ Do not know). Each correct answer will have 1 score, the score ranged from 0 to 10, with higher score indicates better knowledge.
Readiness to quit | From enrolment, 6-week (after treatment) and 12-week follow-up
  To compare the readiness to quit between participants in intervention and control group during the study period using The Contemplation ladder. This measurement is a valid tool consists of 11 rungs ranging from 0 = 'no thought about quitting' to 10 = 'have already quitted', representing 5 stages of change in readiness for cigarette smoking and substance use control.
Attitudes on shisha smoking | From enrolment, 6-week (after treatment) and 12-week follow-up
  To compare the attitudes towards shisha smoking between participants in intervention or control group during the study period by self-designed a 14-item, 5-point Liker scale (ranging from 1 = Strongly disagree to 5 = Strongly agree), the score ranged from 14 to 70, higher score represents more positive attitude towards shisha smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Kai Chun Law, MSc, Principal Investigator — The University of Hong Kong
Locations (1):
- Room 212, New Clinical Building, Queen Mary Hospital, 102 Pokfulam Road, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The dataset without personal identifiers and contact information will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The dataset will be available from May 2026 for 5 years following the principles from the HKSAR Personal Data (Privacy) Ordinance (Cap. 486) and the principles from the Policy on the Management of Research Data and Records, the University of Hong Kong.
Access Criteria: The IPD and supporting information will be available from the PI of this study Mr Law Kai Chun Johnson upon reaonalbe request.
URL: https://stophku.wixsite.com/website

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT07070154/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT07070154/ICF_001.pdf